CLINICAL TRIAL: NCT02083835
Title: Improvement in Postoperative Pain Outcome
Brief Title: PAIN OUT: Improvement in Postoperative PAIN OUTcome
Acronym: PAIN-OUT
Status: Recruiting | Type: Observational
Sponsor: University of Jena (Other)
Collaborators: Jena University Hospital (Other); University of Exeter (Other); University of Leipzig (Other); Region Örebro County (Other); Takwa GmbH (Unknown); University of Basel (Other); Parc de Salut Mar (Other); University Hospital Muenster (Other); Charite University, Berlin, Germany (Other); County Clinical Emergency Hospital Cluj-Napoca (Other); University of London (Other); Luzerner Kantonsspital (Other); Hôpital Raymond Poincaré (Other); Azienda Ospedaliera Santa Maria Degli Angeli (Other); Tel-Aviv Sourasky Medical Center (Other Government); Mälardalens Högskola Västeras (Unknown); University Hospital, Saarland (Other); Insel Gruppe AG, University Hospital Bern (Other); University of Bern (Other); University Hospital, Geneva (Other); University of Lausanne Hospitals (Other); Fox Valley Orthopedic Institute (Other); Landspitali University Hospital (Other); St. Luke's Medical Center (Other); King Hussein Cancer Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Rambam Health Care Campus (Other); Fundación Santa Fe de Bogota (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); Chinese PLA General Hospital (Other); Wuhan TongJi Hospital (Other); University Medical Center Nijmegen (Other); Military Medical Academy, Belgrade, Serbia (Other); Hospital Ambroise Paré Paris (Other); Vrije Universiteit Brussel (Other); Hospital Son Espases (Other); Azienda Ospedaliera (Other); University of Campania Luigi Vanvitelli (Other); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Winfried Meissner, apl. Prof. Dr. med. Winfried Meissner, University of Jena
Other Study IDs: FP7 223590
Record Dates: First submitted 2014-03-03; First posted 2014-03-11 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Post-operative Pain
Keywords: post-operative pain; paitent reported outcomes; quality improvement
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- post-surgical patients: post-surgical patients > 18 years
- pediatric patients post-op day 1: pediatric patients <18 years on post-op day 1 (sub-project QUIPSI - PAIN OUTinfant)

SUMMARY:
PAIN OUT is a multi-national, non-interventional registry and benchmark project, assessing and analysing clinical and patient-reported outcome data of postoperative pain.

DETAILED DESCRIPTION:
PAIN OUT offers a large registry as well as a system for benchmarking and feedback of outcome quality and decision support in acute pain conditions. It collects demographic, clinical and outcome data, using a validated assessment tool available in multiple languages.

The registry part of the project aims at performing population-based research. Furthermore, its infrastructure allows for the conduct of prospective studies comparing the effectiveness of processes of care.

The benchmark part of the project provides the medical community with a unique, user-friendly system to improve treatment of patients with postoperative pain. A web-based information system, featuring two main functions, was developed:

1. a feedback and benchmarking system which provides participating sites with continuously updating data and analyses about the quality of care they provide compared to other institutions and allows identification of best clinical practice.
2. a knowledge library which provides clinicians with easily accessible and regularly updated summaries of evidence-based recommendations tailored to specific post-operative situations.

PAIN OUT is leading and overseeing sub-projects in Mexico, China, a number of European countries. Additional countries will join over time. The sub-projects are scheduled to take place over a period of two years. The design is an uncontrolled pre- post-study, in which approximately 10 hospitals from each country participate. The project consists of collecting data (processes and patient reported outcomes) at baseline from 1-3 wards in participating hospitals; analyzing of the findings, selecting and implementing measures for change in practice; carrying out another round of data collection; summerizing the findings and discussing options for further work.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years or >= 4 years for sub-project QUIPSI/PAIN OUTinfant
* patient is post-op day 1
* patient is at least 6 hours on the ward
* patient has given consent

Exclusion Criteria:

* patient cannot communicate
* patient is cognitively impaired
* patient is asleep
* patient is too ill
* patient does not want to fill in the questionnaire

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adult post-surgical patients in hospitals on post-op day 1
Sampling Method: Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2009-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of postoperative pain treatment | first postoperative day

SECONDARY OUTCOMES:
patients' perception of pain treatment outcome | first postoperative day
  * worst pain since surgery
  * least pain since surgery
  * time in pain
  * interference of pain with activities
  * affect of pain on mood and emotions
  * pain therapy side effects
  * pain relief
  * wish for more treatment
  * information on treatment
  * participation in decisions
  * satisfaction
  * non-medical treatment methods
  * pre-hospital existence of pain

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Meissner, Prof., Study Director — University of Jena
Locations (1):
- Jena University Hospital, Jena, Germany

REFERENCES:
- [Result] Gerbershagen HJ, Pogatzki-Zahn E, Aduckathil S, Peelen LM, Kappen TH, van Wijck AJ, Kalkman CJ, Meissner W. Procedure-specific risk factor analysis for the development of severe postoperative pain. Anesthesiology. 2014 May;120(5):1237-45. doi: 10.1097/ALN.0000000000000108. PMID 24356102
- [Result] Rothaug J, Zaslansky R, Schwenkglenks M, Komann M, Allvin R, Backstrom R, Brill S, Buchholz I, Engel C, Fletcher D, Fodor L, Funk P, Gerbershagen HJ, Gordon DB, Konrad C, Kopf A, Leykin Y, Pogatzki-Zahn E, Puig M, Rawal N, Taylor RS, Ullrich K, Volk T, Yahiaoui-Doktor M, Meissner W. Patients' perception of postoperative pain management: validation of the International Pain Outcomes (IPO) questionnaire. J Pain. 2013 Nov;14(11):1361-70. doi: 10.1016/j.jpain.2013.05.016. Epub 2013 Sep 7. PMID 24021577
- [Result] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Result] Gerbershagen HJ, Rothaug J, Kalkman CJ, Meissner W. Determination of moderate-to-severe postoperative pain on the numeric rating scale: a cut-off point analysis applying four different methods. Br J Anaesth. 2011 Oct;107(4):619-26. doi: 10.1093/bja/aer195. Epub 2011 Jun 30. PMID 21724620
- [Result] Rothaug J, Weiss T, Meissner W. How simple can it get? Measuring pain with NRS items or binary items. Clin J Pain. 2013 Mar;29(3):224-32. doi: 10.1097/AJP.0b013e31824c5d7a. PMID 23369928
- [Result] Taylor RS, Ullrich K, Regan S, Broussard C, Schwenkglenks M, Taylor RJ, Gordon DB, Zaslansky R, Meissner W, Rothaug J, Langford R; PAIN-OUT investigators. The impact of early postoperative pain on health-related quality of life. Pain Pract. 2013 Sep;13(7):515-23. doi: 10.1111/papr.12026. Epub 2012 Dec 23. PMID 23279591
- [Result] Zaslansky R, Chapman CR, Rothaug J, Backstrom R, Brill S, Davidson E, Elessi K, Fletcher D, Fodor L, Karanja E, Konrad C, Kopf A, Leykin Y, Lipman A, Puig M, Rawal N, Schug S, Ullrich K, Volk T, Meissner W. Feasibility of international data collection and feedback on post-operative pain data: proof of concept. Eur J Pain. 2012 Mar;16(3):430-8. doi: 10.1002/j.1532-2149.2011.00024.x. Epub 2011 Dec 19. PMID 22337250
- [Result] Zaslansky R, Rothaug J, Chapman CR, Backstrom R, Brill S, Fletcher D, Fodor L, Gordon DB, Komann M, Konrad C, Leykin Y, Pogatski-Zahn E, Puig MM, Rawal N, Ullrich K, Volk T, Meissner W. PAIN OUT: the making of an international acute pain registry. Eur J Pain. 2015 Apr;19(4):490-502. doi: 10.1002/ejp.571. Epub 2014 Aug 12. PMID 25132607
- [Result] Zaslansky R, Rothaug J, Chapman RC, Backstrom R, Brill S, Engel C, Fletcher D, Fodor L, Funk P, Gordon D, Komann M, Konrad C, Kopf A, Leykin Y, Pogatzki-Zahn E, Puig M, Rawal N, Schwenkglenks M, Taylor RS, Ullrich K, Volk T, Yahiaoui-Doktor M, Meissner W. PAIN OUT: an international acute pain registry supporting clinicians in decision making and in quality improvement activities. J Eval Clin Pract. 2014 Dec;20(6):1090-8. doi: 10.1111/jep.12205. Epub 2014 Jul 1. PMID 24986116
- [Result] Polanco-Garcia M, Garcia-Lopez J, Fabregas N, Meissner W, Puig MM; PAIN-OUT-Spain Consortium. Postoperative Pain Management in Spanish Hospitals: A Cohort Study Using the PAIN-OUT Registry. J Pain. 2017 Oct;18(10):1237-1252. doi: 10.1016/j.jpain.2017.05.006. Epub 2017 Jun 12. PMID 28619696
- [Result] Komann M, Weinmann C, Schwenkglenks M, Meissner W. Non-Pharmacological Methods and Post-Operative Pain Relief: An Observational Study. Anesth Pain Med. 2019 Apr 20;9(2):e84674. doi: 10.5812/aapm.84674. eCollection 2019 Apr. PMID 31341822
- [Result] Dubljanin Raspopovic E, Meissner W, Zaslansky R, Kadija M, Tomanovic Vujadinovic S, Tulic G. Associations between early postoperative pain outcome measures and late functional outcomes in patients after knee arthroplasty. PLoS One. 2021 Jul 28;16(7):e0253147. doi: 10.1371/journal.pone.0253147. eCollection 2021. PMID 34320012
- [Result] Garduno-Lopez AL, Acosta Nava VM, Castro Garces L, Rascon-Martinez DM, Cuellar-Guzman LF, Flores-Villanueva ME, Villegas-Sotelo E, Carrillo-Torres O, Vilchis-Samano H, Calderon-Vidal M, Islas-Lagunas G, Richard Chapman C, Komann M, Meissner W, Baumbach P, Zaslansky R. Towards Better Perioperative Pain Management in Mexico: A Study in a Network of Hospitals Using Quality Improvement Methods from PAIN OUT. J Pain Res. 2021 Feb 15;14:415-430. doi: 10.2147/JPR.S282850. eCollection 2021. PMID 33623424
- [Result] van Dijk JFM, Zaslansky R, van Boekel RLM, Cheuk-Alam JM, Baart SJ, Huygen FJPM, Rijsdijk M. Postoperative Pain and Age: A Retrospective Cohort Association Study. Anesthesiology. 2021 Dec 1;135(6):1104-1119. doi: 10.1097/ALN.0000000000004000. PMID 34731245
- [Result] van Driel MEC, van Dijk JFM, Baart SJ, Meissner W, Huygen FJPM, Rijsdijk M. Development and validation of a multivariable prediction model for early prediction of chronic postsurgical pain in adults: a prospective cohort study. Br J Anaesth. 2022 Sep;129(3):407-415. doi: 10.1016/j.bja.2022.04.030. Epub 2022 Jun 19. PMID 35732539
- [Result] Hofer DM, Lehmann T, Zaslansky R, Harnik M, Meissner W, Stuber F, Stamer UM. Rethinking the definition of chronic postsurgical pain: composites of patient-reported pain-related outcomes vs pain intensities alone. Pain. 2022 Dec 1;163(12):2457-2465. doi: 10.1097/j.pain.0000000000002653. Epub 2022 Apr 19. PMID 35442934
- [Derived] Harnik MA, Oswald O, Huber M, Hofer DM, Komann M, Dreiling J, Stamer UM. Multidimensional pain assessment and opioid use after total knee arthroplasty: continuous vs single-injection regional vs systemic analgesia. Pain Rep. 2025 Mar 18;10(2):e1257. doi: 10.1097/PR9.0000000000001257. eCollection 2025 Apr. PMID 40109369
- [Derived] Hofer DM, Harnik M, Lehmann T, Stuber F, Baumbach P, Dreiling J, Meissner W, Stamer UM. Trajectories of pain and opioid use up to one year after surgery: analysis of a European registry. Br J Anaesth. 2024 Mar;132(3):588-598. doi: 10.1016/j.bja.2023.12.002. Epub 2024 Jan 10. PMID 38212183
- [Derived] Bernhart K, Becke-Jakob K, Lehmann T, Harnik M, Seiler S, Meissner W, Stuber F, Stamer UM. Analgesic use and favourable patient-reported outcome measures after paediatric surgery: an analysis of registry data. Br J Anaesth. 2023 Jan;130(1):74-82. doi: 10.1016/j.bja.2022.09.028. Epub 2022 Dec 5. PMID 36470745
- [Derived] Jiang B, Wu Y, Wang X, Gan Y, Wei P, Mi W, Feng Y. The influence of involving patients in postoperative pain treatment decisions on pain-related patient-reported outcomes: A STROBE-compliant registering observational study. Medicine (Baltimore). 2022 Sep 23;101(38):e30727. doi: 10.1097/MD.0000000000030727. PMID 36197159
- [Derived] Polanco-Garcia M, Granero R, Gallart L, Garcia-Lopez J, Montes A. Finding the vulnerable postoperative population: A two-step cluster analysis of the PAIN-OUT registry. Eur J Pain. 2022 Sep;26(8):1732-1745. doi: 10.1002/ejp.1997. Epub 2022 Jul 7. PMID 35762292
- [Derived] Zaslansky R, Meissner W, Chapman CR. Pain after orthopaedic surgery: differences in patient reported outcomes in the United States vs internationally. An observational study from the PAIN OUT dataset. Br J Anaesth. 2018 Apr;120(4):790-797. doi: 10.1016/j.bja.2017.11.109. Epub 2018 Feb 2. PMID 29576119
- [Derived] Stamer UM, Naef N, Porz R, Stuber F, Leva B, Meissner W, Fletcher D; euCPSP Study Group. Ethical procedures and patient consent differ in Europe. Eur J Anaesthesiol. 2015 Feb;32(2):126-31. doi: 10.1097/EJA.0000000000000206. PMID 25503525
- See also: Project webpage — http://www.pain-out.eu